CLINICAL TRIAL: NCT01864538
Title: A Phase 2 Biomarker - Enriched Study of TH-302 in Subjects With Advanced Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: ImmunoGenesis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-413
Record Dates: First submitted 2013-05-13; First posted 2013-05-29 (Estimated); Results first posted 2017-08-16 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Melanoma
Keywords: TH-302; Advanced Melanoma; Metastatic; Biomarker; Mucosal Melanoma; Evofosfamide
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — TH 302

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TH-302 (Experimental): 480 mg/m2 by iv infusion over 30 - 60 min on Days 1, 8, and 15 of a 28-day cycle.
  Interventions: Drug: TH-302

INTERVENTIONS:
Drug: TH-302 — 480 mg/m2 by iv infusion over 30 - 60 min on Days 1, 8, and 15 of a 28-day cycle.

SUMMARY:
The primary objective of this study is to determine the response rate, duration of response,progression-free survival and overall survival of subjects with advanced melanoma treated with TH-302.

DETAILED DESCRIPTION:
Hypoxia is an independent marker of a poor prognosis for subjects with metastatic melanoma (Simonetti 2012, Lartigau 1997). Hypoxic melanoma cells are more likely to exhibit a stem-cell like phenotype with an associated increased propensity for invasion, angiogenesis, and metastasis formation compared to normoxic cells. Moreover, this phenotype is also associated with treatment resistance. TH-302, a hypoxia activated prodrug (HAP), was designed to target the hypoxic nature of tumours while having a minimal effect on normoxic tissue. TH-302 belongs to a class of alkylating agents that have significant experimental and clinical activity (Brock 1989). Preclinical data support the hypothesis that TH-302 targets hypoxic regions of tumours and is also able to kill tumour cells in normoxic regions as a result of cytotoxin diffusion, leading to significant effects on tumour growth (Meng 2011). TH-302 has been investigated in over 700 subjects with solid tumours or hematologic malignancies, including subjects with metastatic melanoma. In this subset a disease control rate of 63% (3 subjects with partial responses and 9 subjects with stable disease out of a total of 19) was observed in an early phase clinical trial of TH-302 (Weber 2010). Predictive biomarkers for response and toxicity have yet to be identified for subjects with advanced melanoma treated with TH-302. Optimal patient selection may be critical to maximize the clinical benefit. A predictive biomarker approach will be investigated to try to identify subjects most likely to benefit from TH-302. Given the hypoxia-targeting mechanism of TH- 302, it is believed that hypoxia biomarkers will be the most informative for identifying subjects likely to benefit from TH- 302; however, additional biomarkers including DNA repair biomarkers will also be investigated. In addition, this approach will also have potential to synergise with future immunotherapeutic approaches as suppressive T regulatory cells are thought to reside within hypoxic niches within the tumour microenvironment that would be amenable to targeting by TH-302.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's Regional Ethics Board/Independent Ethics Committee (REB/IEC)
3. Histologically documented cutaneous or mucosal malignant melanoma, which is recurrent or metastatic and is not curable by surgical or other means.
4. Adequate tumour tissue (greater than 0.5cm3 preferred, 3 X core biopsy acceptable) available and agreement from subjects that this tissue from their primary and/or metastatic tumour be made available for assessment of potential biomarkers.
5. Ability and availability to complete all prescribed biomarker studies (Screening and after Cycle 2).
6. Recovered to Grade 1 from reversible toxicities of prior therapy
7. Presence of clinically and/or radiologically documented disease. At least one site of disease (which will not be removed during the course of the study) must be uni-dimensionally measurable as per RECIST 1.1 or clinically quantifiable (such as in the case of skin disease)
8. ECOG performance status of 0 - 1.
9. Prior treatment with any number of immunotherapies (e.g., IL2, ipilimumab), targeted therapies (e.g., vemurafenib) are permitted but no more than one 1 prior chemotherapy
10. Acceptable liver function
11. Acceptable renal function
12. Acceptable hematologic status (without growth factor support for neutropenia or transfusion dependency):
13. Normal 12-lead ECG (clinically insignificant abnormalities permitted)
14. Female subjects of childbearing age must have a negative urine HCG test unless prior hysterectomy or menopause (defined as age above 55 and twelve months without menstrual activity). Female subjects should not become pregnant or breast-feed while on this study. Sexually active male and female subjects should use effective birth control.

Exclusion Criteria:

1. Anticancer treatment with radiation therapy, targeted therapies, chemotherapy, immunotherapy, hormones or other antitumour therapies within 28 days prior to first dose of TH-302.
2. Subjects who have received any other investigational drug or agent within 28 days of first dose of TH-302
3. Current use of drugs with known cardiotoxicity
4. Significant cardiac dysfunction:
5. Seizure disorders requiring anticonvulsant therapy
6. Progressing brain metastases (unless previously treated and stable disease for a period of greater than or equal to 3 months on repeat MRI following definitive treatment).
7. History of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for greater than 2 years
8. Severe chronic obstructive or other pulmonary disease with hypoxemia (requires supplementary oxygen, symptoms due to hypoxemia or oxygen saturation less than 90% by pulse oximetry after a 2 minute walk) or in the opinion of the investigator any physiological state likely to cause hypoxia of normal tissue.
9. Major surgery, other than diagnostic surgery, within 4 weeks prior to Cycle 1 Day 1, without complete recovery
10. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
11. Prior therapy with an hypoxic cytotoxin
12. Known infection with HIV or active infection with hepatitis B or hepatitis C
13. History of allergic reaction to a structural compound or biological agent similar to TH-302
14. Pregnancy or breast-feeding
15. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
16. Unwillingness or inability to comply with the study protocol for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tillman Pearce, MD, Study Director — Threshold Pharmaceuticals
Locations (7):
- United States (3):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - UCLA, Los Angeles, California
  - Columbia University Medical Center, New York, New York
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TH-302
Started | 11
Completed | 0
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | TH-302
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | TH-302
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Arm/Group | TH-302
Serious Adverse Events (participants affected / at risk) | 8/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TH-302 (N=11)
Cellulitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Splenic thrombosis (Blood and lymphatic system disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TH-302 (N=11)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 3 (5)
Vomiting (Gastrointestinal disorders) | 2 (4)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2)
Chills (General disorders) | 2 (3)
Fatigue (General disorders) | 6 (10)
Oedema peripheral (General disorders) | 4 (4)
Pyrexia (General disorders) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Weight decreased (Investigations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No